CLINICAL TRIAL: NCT00251069
Title: Glucosamine Sulphate and Hypercholesterolaemia
Brief Title: Glucosamine Sulphate and Increased Level of Blood Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Slidgigtinstituttet (Other)
Collaborators: Pharma Nord (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCTnr 2005-000541-11
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2005-11-09 (Estimated); Status verified 2005-07

CONDITIONS: Osteoarthritis
Keywords: glucosamine sulphate, osteoarthritis, cholesterol,
MeSH Terms: conditions — Osteoarthritis | interventions — Glucosamine

INTERVENTIONS:
Drug: Glucosamine sulphate

SUMMARY:
Glucosamine sulphate causes no changes in blood levels of cholesterol

DETAILED DESCRIPTION:
The effects on glucosamine sulphate on blood levels of choleterol is measuered in patients with mild to moderate osteoarthritis

ELIGIBILITY:
Inclusion Criteria: Osteoarthritic pain, normal blood cholesterol levels -

Exclusion Criteria: Systemic diseases, pregnancy, need of medication besides painkillers

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2005-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Levels of blood cholesterol

SECONDARY OUTCOMES:
Effect of treatment on pain

CONTACTS AND LOCATIONS:
Overall Officials: Keld Ostergaard, M.D., Ph.D., Principal Investigator — Slidgigtinstituttet
Locations (1):
- Slidgigtinstituttet, Ishøj, Denmark